CLINICAL TRIAL: NCT02160444
Title: Investigating the Effects of an Added Parent Component to Cognitive Behavior Therapy for Youth With Anxiety Disorders
Brief Title: Investigating the Effects of Parent Component to Cognitive Behavior Therapy (CBT) for Youth With Anxiety Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Kevin D. Stark, Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-05-0009
Record Dates: First submitted 2013-07-14; First posted 2014-06-10 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Anxiety Disorders
Keywords: CBT; Parent Training; Anxiety Disorders in Children
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT plus Parent as CBT Coach Training (Experimental): CBT plus Parent as CBT Coach Training
  Interventions: Behavioral: CBT plus Parent as CBT Coach Training

INTERVENTIONS:
Behavioral: CBT plus Parent as CBT Coach Training — Standard CBT for treatment of anxiety disorders in youth is completed by the children while their primary caregiver receives training in the same cognitive behavioral skills, how to recognize when he or she is accommodating his or her child's anxiety, and how to create and implement exposure activities.

SUMMARY:
Investigation is designed to determine whether the gold standard for treating anxious youth is enhanced by teaching parents to become their anxious child's CBT coach. Children (7-17 years old) with either Generalized Anxiety Disorder, Social Phobia, or Separation Anxiety Disorder are treated with a combination of the Coping Cat Program and a parent-training intervention that is designed to teach the child's parents the same cognitive and behavioral skills that the child is learning and how to help their child to complete exposure activities. The research methods are parallel to those used in the CAMS study so that this data can be merged with that data set to evaluate the relative efficacy of the enhanced intervention.

DETAILED DESCRIPTION:
Children between the ages of 7 and 17 years old who are primarily experiencing either Generalized Anxiety Disorder, Separation Anxiety Disorder or Social Phobia and are not experiencing a cognitive or learning disability that would prevent them from validly completing the measures are eligible for participation in the study. Children who are experiencing another psychological disorder as their primary disorder would be excluded from the current investigation. Outcome measures include the ADIS for Diagnostic and Statistical Manual (fourth edition)(DSM-IV( Child or Parent, Children's Global Improvement Scale (CGI-I), Children's Global Assessment Scale (CGAS), Pediatric Anxiety Rating Scale (PARS), Negative Affect Self-Statements Questionnaire (NASSQ), Coping Questionnaire (CQ), Goal Attainment Scale (GAS), Mood and Feelings Questionnaire (MFQ), Multi-dimensional Anxiety Scale for Children (MASC), Screen for Child Anxiety and Related Emotional Disorders (SCARED),Family Assessment Measure (third editions) (FAM-III Dyadic), Perception of Therapeutic Relationship (PTR), Satisfaction Questionnaire (SQ), Child Behavior Check List (CBCL), Family Burden Assessment Scale (BAS), Brief Symptom Index (BSI), State Trait Anxiety Inventory (STAI), Brief Family Assessment Measure (third editions (Brief FAM-III).

ELIGIBILITY:
Inclusion Criteria:

* Child is between 7-17 years old
* Primary diagnosis of Generalized Anxiety Disorder
* Separation Anxiety Disorder, or Social Phobia.

Exclusion Criteria:

* Presence of Major Depression, suicidal risk, presence of a learning disability or cognitive deficit that would prevent the child from validly completing the measures
* Presence of another psychological disorder that is of primary significance

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2012-06; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale measures change in severity of anxiety from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Interview measure of the severity of anxiety symptoms that is completed by the child and his or her primary caregiver.
Multidimensional Anxiety Scale for Children measures change in severity of anxiety from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of severity of anxiety symptoms in children and adolescents.
Screen for Child Anxiety Related Emotional Disorders measures change in severity of anxiety and related co-morbid disorders from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of the severity of anxiety symptoms.
Clinical Global Severity and Improvement Scales measure change in severity of anxiety and co-morbid disorders from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assessment of initial severity of illness and extent of improvement over treatment and follow-ups.
Children's Global Assessment Scale measures change in severity of anxiety and co-morbid disorders from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assessment of the degree of overall functioning of the child participants.
Anxiety Disorders Schedule for DSM-IV: Child Version and Parent Version | Baseline(One week prior to starting treatment)
  Interview measure of the presence and severity of various anxiety disorders and common co-existing disorders.

SECONDARY OUTCOMES:
Family Assessment Measure III, Dyadic Relationship Scale measures change in perceived family environment from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assess family relationships
Child Behavior Checklist measures change in severity of internalizing and externalizing symptoms from the parent's perspective from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Broadband measure of child psychopathology
Family Burden Assessment measures change in severity of the burden the child's anxiety disorder creates for the family from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of the impact on the family of the child's anxiety disorder.
Brief Symptom Inventory measures change in severity of parental psychopathology from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assess parental psychopathology
State Trait Anxiety Inventory measures change in severity of anxiety for parents from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measures anxiety symptoms in parents.
Mood and Feelings Questionnaire measures change in severity of depressive symptoms from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of depressive symptoms in the child participants
Goal Attainment Scale measures goal attainment from baseline to post-treatment and assess maintenance of goal attainment at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Therapist sets five goals for the child patient and then tracks progress over the course of treatment.
Coping Questionnaire measures change in coping skills from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assess for the presence of coping skills in the child participants.
Negative Affective Self-Statement Questionnaire measures change in negative cognitions from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of negative cognitions in the child participants.
Harm to Self and Others Interview measures change in suicidal ideation, homicidal ideation and self-harming behaviors from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assessment of suicidal, homicidal and self-harm behavior and ideation.

OTHER OUTCOMES:
Perception of Therapeutic Relationship measures the participants' satisfaction with the therapeutic relationship at post-treatment and at the one year and two year follow-ups. | Post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assesses the patient-therapist relationship from the patient's perspective.
Satisfaction Questionnaire measures the degree of satisfaction the participants experience at post-treatment and at one and two year follow-up assessments. | Post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assesses the extent to which the patients are satisfied with the treatment they received.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D. Stark, Ph.D., Principal Investigator — University of Texas
Locations (1):
- Texas Child Study Center, Austin, Texas, United States

REFERENCES:
- See also: Link for the Texas Child Study Center — http://www.dellchildrens.net/services_and_programs/texas_child_study_center__mental_health_services/